CLINICAL TRIAL: NCT04248660
Title: Comparison of Uterine Artery Doppler Measurements Performed at 11-14 and 20-22 Weeks of Gestation During Pregnancy According to Delivery Type and Number of Births and Investigation of the Effects on Obstetric Outcomes (Maternal, Fetal, Neonatal Results)
Brief Title: Uterine Artery Doppler and 11-14 / 20-22 Weeks of Gestation Pregnancy
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, Pınar kadirogullari, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: ATADEK-2020/00
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Pregnancy Related
Keywords: Uterine artery doppler; type of delivery; obstetric outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uterine artery doppler measurements: Uterine artery doppler measurements will be made in the same patients at 11-14 weeks and 20-22 weeks of pregnancy.
  Doppler results will be classified according to pregnancy results and primary results will be doppler findings.
  Interventions: Other: uterine artery doppler measurement

INTERVENTIONS:
Other: uterine artery doppler measurement — The effect of delivery type on changes in uterine blood flow will be investigated.
  Doppler results groups will be defined according to the effect of deviations in uterine blood flow on neonatal and perinatal results.

SUMMARY:
Uterine artery doppler measurements will be made at 11-14 weeks and 20-22 weeks of gestation, and the classification of these measurements according to type of delivery; and to investigate the change in the effect of delivery type on uterine artery flows on obstetric outcomes (maternal, fetal, neonatal outcomes).

DETAILED DESCRIPTION:
The first and second trimester perinatal examination results performed by the same operator from pregnant women who have applied to the clinic since the first trimester are removed from the ViewPoint 6.0 server and database and their uterine artery doppler values (uterine artery PI and RI values, presence of uterine artery notch), placental location, gestational week of measurement, blood pressures, PAPP-A and hCG MoM values, obstetric results (type of birth, week, weight, ante-postpartum complications), data to be generated from other hospital records will be saved to the base

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 11-14. applying to the outpatient clinic at week
* Single spontaneous pregnancy
* Having a first pregnancy (primigravid nullipar) or having given birth once (primipar) (first birth by vaginal route or cesarean)
* Result of previous pregnancy with live birth (term delivery without obstetric complication)
* No intrauterine growth restriction in the first pregnancy
* Women who gave birth by cesarean section were not placed due to caesarean indication due to placental location-invasion anomaly, maternal chronic disease (hypertension, diabetes, coronary artery disease, etc.), placental detachment.

Exclusion Criteria:

* Multiple pregnancies
* Pregnancies with assisted reproductive techniques
* Placental anomaly in previous pregnancy
* Maternal chronic hypertension, preeclampsia, history of diabetes
* Pregnant women who smoke
* The presence of fetal chromosomal or structural anomaly
* two or more cesarean sections
* Having undergone non-cesarean surgery (myomectomy, septum or polyp resection ... etc)
* Presence of uterine structural anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who had uterine artery doppler measurements and delivered at 11-14 weeks and 20-22 weeks of pregnancy will be the study group. these patients; Doppler results will be classified according to pregnancy results, and the classification of these measurements according to type of delivery; and the effect of delivery on uterine artery flows on obstetric outcomes (maternal, fetal, neonatal outcomes) will be examined.
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Doppler results of 11-14 weeks of gestation in patients with previous cesarean section | 10 months
  uterine artery doppler values (uterine artery PI , presence of uterine artery notch)
Doppler results of 11-14 weeks of gestation in those who gave birth beforehand | 10 months
  uterine artery doppler values (uterine artery PI , presence of uterine artery notch)
Doppler results of 20-22 weeks of gestation in patients with previous cesarean section | 10 months
  uterine artery doppler values (uterine artery PI , presence of uterine artery notch)
Doppler results of 20-22 weeks of gestation in those who gave birth beforehand | 10 months
  uterine artery doppler values (uterine artery PI , presence of uterine artery notch)

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)